CLINICAL TRIAL: NCT01884428
Title: Phase I, Prospective, Open-label, Multi-centric, Dose Finding Trial of Combination of IGEV and Panobinostat Before Autologous Stem Cell Transplant in Patients With Hodgkin's Lymphoma
Brief Title: Study of Combination of PIGEV Before Autologous Stem Cell Transplant in Patients With Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, MD, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2010-003; 2010-022452-23 (EudraCT Number)
Record Dates: First submitted 2013-05-27; First posted 2013-06-24 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin; Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — Panobinostat; Ifosfamide; Gemcitabine; Vinorelbine; Prednisolone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panobinostat + IGEV (Experimental): Panobinostat + IGEV regimen (Ifosfamide, Gemcitabine, Vinorelbine, Prednisolone)
  Interventions: Drug: panobinostat; Drug: Ifosfamide; Drug: Gemcitabine; Drug: Vinorelbine; Drug: Prednisolone

INTERVENTIONS:
Drug: panobinostat — Dose excalation oral panobinostat 3 days a week for a maximum of 4 cycles of three weeks duration
  Other Names: LBH-589
Drug: Ifosfamide — Ifosfamide 2000 mg/m2 on days 1 to 4 as a 2-hour infusion for a maximum of 4 cycles of three weeks duration
  Other Names: Ifex
Drug: Gemcitabine — Gemcitabine 800 mg/m2 on days 1 and 4 for a maximum of 4 cycles of three weeks duration
  Other Names: Gemzar
Drug: Vinorelbine — Vinorelbine 20 mg/m2 on day 1 for a maximum of 4 cycles of three weeks duration
  Other Names: Navelbine
Drug: Prednisolone — Prednisolone 100 mg on days 1 to 4 for a maximum of 4 cycles of three weeks duration
  Other Names: Prelone

SUMMARY:
study to assess maximum tolerated dose (MTD), safety, tolerability and activity of IGEV (Ifosfamide, Gemcitabine,Vinorelbine, Prednisolone) + Panobinostat new combination in order to determine the recommended phase II dose

DETAILED DESCRIPTION:
Patients will received 4 p-IGEV courses repeated every 3 weeks in the absence of unacceptable toxicity, whenever an objective response is observed at disease evaluation performed after II cycle.

Eligible patients will be accrued in cohorts of 3 patients at each dose level and dose escalation will be performed following the standard 3+3 rule.

Three patients will be treated for each dose-level, starting from level 1, for one cycle: if no dose-limiting toxicities (DLTs) will be recorded after the first cycle, treatment will be continued in those patients until study completion or unacceptable toxicity and three new patients will be treated at the next dose level. However, if one out of 3 patients will develop a DLT, the same dose-level will be administered to three additional patients for one cycle. If no one of those additional patients will experience a DLT, dose escalation will continue. If more than one over 3 or 6 patients will develop a DLT after the first cycle in any cohort, MTD will be reached. Six further patients will be treated at the lower dose in order to obtain more information about the optimal dose for phase II trials and to characterize pharmacokinetic profiles of this combination. If DLT will be found at level 1 (20 mg), 3 patients will be treated at dose -1 (10 mg). If no more than 1 patient experience toxicity, other 3 patients will be treated to assess more information about pharmacokinetic profiles and safety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed or refractory classical HL
* Measurable disease
* One or two prior systemic lines of treatment
* PS(ECOG) 0-2
* Absence of bone marrow infiltration
* Adequate laboratory values for bone marrow, liver and renal functionality

Exclusion Criteria:

* prior or concurrent treatment with a DAC inhibitor including panobinostat
* valproic acid therapy for any medical condition during the study or within 5 days prior to the first panobinostat treatment
* previous autologous hematopoietic stem cell transplant
* other concurrent therapy intended to treat the primary cancer including chemotherapy, investigational or biologic agents or other antitumor agents
* impaired cardiac function or unstable AF
* known history of HIV seropositivity, chronic hepatitis, or other active viral infections
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of panobinostat (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, obstruction, or stomach and/or small bowel resection)
* pregnant or breast feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-03 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) or the recommended phase II dose defined as the highest dosage cohort at which no more than one of six patients will experience a DLT in the first treatment cycle. | 3 weeks

SECONDARY OUTCOMES:
DLT | 3 weeks
  Incidence of dose limiting toxicities (DLTs)
safety profile | 3 months
  Preliminary safety profile defined as Adverse Events (AEs), Serious Adverse Events ( SAEs) & Changes in Clinical Laboratory Evaluations
Complete Response and Overall Response Rate | 3 months
hematologic toxicity | 3 months
  Assessment of neutropenia and thrombocytopenia incidence, duration, as well as platelet transfusion requirement
CD34+ cells count | 3 months
  Assessment of number of CD34+ collected and number of leukapheresis required to obtain an appropriate collection according to transplant program.
efficacy of PIGEV combination in terms of progression-free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Italy